CLINICAL TRIAL: NCT00005852
Title: Allogeneic Bone Marrow Transplantation for Marrow Failure States
Brief Title: Bone Marrow Transplantation in Treating Patients With Severe Aplastic Anemia or Rejection of Previous Bone Marrow Transplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: MCC-11309; MCC-11309; MCC-IRB-4251; NCI-G00-1791
Record Dates: First submitted 2000-06-02; First posted 2004-07-26 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Myeloproliferative Disorders; Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; primary myelofibrosis; childhood acute promyelocytic leukemia (M3); refractory hairy cell leukemia; recurrent/refractory childhood Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; graft versus host disease; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Primary Myelofibrosis; Leukemia, Hairy Cell; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Antilymphocyte Serum; Filgrastim; Muromonab-CD3; Cyclophosphamide; Cyclosporine; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: filgrastim
Biological: muromonab-CD3
Drug: cyclophosphamide
Drug: cyclosporine
Drug: methylprednisolone
Procedure: allogeneic bone marrow transplantation

SUMMARY:
RATIONALE: Bone marrow from donors may be able to treat patients with severe aplastic anemia and patients whose bodies have rejected previous bone marrow transplantation.

PURPOSE: Phase II trial to study the effectiveness of bone marrow transplantation in treating patients who have severe aplastic anemia or whose bodies have rejected previous bone marrow transplant.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the graft failure rate and overall survival of patients with severe aplastic anemia after receiving an allogeneic bone marrow transplant. II. Determine the efficacy of high dose cyclophosphamide and antithymocyte globulin as conditioning regimen for a second bone marrow transplant in patients who reject their first graft. III. Determine the efficacy of methylprednisolone and anti-CD3 monoclonal antibody as a conditioning regimen for a second bone marrow transplant in patients who reject their first graft and are poor candidates for cyclophosphamide and antithymocyte globulin.

OUTLINE: Patients with graft failure with the following organ function and performance status are assigned to arm I: Performance status: Karnofsky 60-100% Pulmonary: FEV1 and DLCO at least 50% Cardiac: Left ventricular ejection fraction at least 45% Hepatic: None to mild venoocclusive disease Patients with graft failure with the following organ function and performance status are assigned to arm II: Performance status: Karnofsky 20-50% Pulmonary: FEV1 or DLCO less than 50% Cardiac: Left ventricular ejection fraction less than 45% Hepatic: Moderate to severe venoocclusive disease Patients with aplastic anemia are assigned to arm I. Arm I: Patients receive cyclophosphamide IV over 1 hour on days -5 to -2, antithymocyte globulin IV over 8 hours on days -5 to -3, and bone marrow transplant on day 0. Arm II: Patients receive methylprednisolone IV twice a day on days -5 to 62; monoclonal antibody OKT3 IV on days -1 to 24; bone marrow transplant on day 0; oral cyclosporine twice a day starting day 20; and filgrastim (G-CSF) subcutaneously once a day starting day -5 until blood counts recover. Patients are followed once a week for 3 months and then monthly for one year.

PROJECTED ACCRUAL: A total of 40 patients (20 with aplastic anemia and 20 with graft failure) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed aplastic anemia Must have related donor with a genotypic 6 out of 6 HLA A, B, and DR match OR Bone marrow transplant failure Must have related donor with at least a 5 out of 6 HLA match OR Must have an unrelated donor with at least a 5 out of 6 HLA match

PATIENT CHARACTERISTICS: Age: 15 to 55 Performance status: Aplastic anemia patients: Karnofsky 80-100% Graft failure patients: Karnofsky 20-100% Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: Aplastic anemia patients: Bilirubin no greater than 2.0 mg/dL SGOT/SGPT no greater than 3 times normal PT/PTT normal (except when aplastic anemia secondary to viral hepatitis) Graft failure patients: Mild to severe venoocclusive disease allowed Renal: Aplastic anemia patients: Creatinine no greater than 2.0 mg/dL Creatinine clearance at least 60 mL/min Cardiovascular: Aplastic anemia patients: Left ventricular ejection fraction at least 45% by MUGA or echocardiography No myocardial infarction within the past 6 months No uncontrolled arrhythmias Pulmonary: Aplastic anemia patients: FEV1 and DLCO at least 50% predicted Other: Aplastic anemia patients: No uncontrolled diabetes mellitus or thyroid disease No active serious infections HIV negative Not pregnant or nursing Negative pregnancy test No psychosocial problem that would preclude study compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1996-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven C. Goldstein, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute